CLINICAL TRIAL: NCT01933698
Title: Bioequivalence Study of Two Commercial Amoxicillin Suspension Formulations in Healthy Human Volunteers
Brief Title: Bioequivalence of Two Commercial Amoxicillin Suspensions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Stiefel, a GSK Company (Industry)
Responsible Party: Principal Investigator, Francisco Groppo, Full Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AMOXIPED-01; 63.064.653/0001-54 (Other Grant/Funding Number: LABORATÓRIOS STIEFEL LTDA)
Record Dates: First submitted 2013-08-20; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Bioequivalence of Amoxicillin
Keywords: Bioequivalence; Amoxicillin; Human
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxi-Ped (Active Comparator): Single dose of 500 mg amoxicillin - AMOXI-PED - was administered after a 12-hour overnight fast.
  Interventions: Drug: amoxicillin
- Amoxil (Active Comparator): Single dose of 500 mg amoxicillin - AMOXIL - was administered after a 12-hour overnight fast.
  Interventions: Drug: amoxicillin

INTERVENTIONS:
Drug: amoxicillin — Comparison of pharmacokinetics of both formulations
  Other Names: Amoxil; Amoxi-Ped

SUMMARY:
The aim of the present study was to compare the pharmacokinetic profiles and to evaluate the bioequivalence of two commercial amoxicillin-suspension formulations in healthy Brazilian volunteers.

DETAILED DESCRIPTION:
Under fasting condition, 25 volunteers (13 males and 12 females) were included in this randomized, open-label, two-period crossover (1-week washout interval) bioequivalence study. Blood samples were collected at pre-dose (0h) and 0.5, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8 and 12 hours after drug ingestion. Pharmacokinetic parameters (Cmax, Tmax, T1/2, Area-under-curve0-12h and Area-under-curve0-inf) were calculated from plasma concentrations for both formulations in each subject.

ELIGIBILITY:
Inclusion Criteria:

* negative to HIV, hepatitis B virus, hepatitis C virus, addictive drugs and pregnancy test for women
* age between 19 and 46 years
* weight between 52 and 85 kg and body mass index between 17.6 and 28.4kg/m2
* ability to provide written consent
* laboratory exam results within the normal range for healthy individuals and/or medically acceptable defined by a clinical investigator;
* feeding habits consistent with the standardization of the study

Exclusion Criteria:

* pregnancy
* history of hypersensitivity to penicillins (normal or idiosyncratic drug reaction)
* any evidence of dysfunction or clinically significant deviation from normal
* history of any psychiatric illness that might compromise the ability to provide written consent
* history of gastrointestinal disease, hepatic, renal, pulmonary, cardiovascular, hematological, neurological or diabetes or glaucoma
* active smoker
* consumption of more than 5 cups of coffee or tea per day
* history of drug dependence or abuse of alcohol consumption
* use of enzymatic-inducers drugs within 30 days or any systemic medication (including prescription drugs, such as painkillers, hepatoprotective, influenza, etc) within 14 days before the start of the study
* participation in any clinical study in 9 weeks prior to the study
* have lost or donated more than 350 mL of blood in the last three months
* have been subjected to abnormal diet for any reason (therapeutic, aesthetic, religious, etc.)
* did not have adequate venous access.

Ages: 19 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2005-02; Primary Completion 2005-05 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Changes in plasmatic amoxicillin concentrations along time measured by HPLC. | Change from baseline to 12 hours
  Amoxicillin were extracted from plasma by precipitating plasma proteins with acetonitrile. Amoxicillin plasmatic concentration was accessed every 30 minutes until 3h hours after drug administration and every 2h after this time until 12h of drug administration. Drug plasmatic concentrations were obtained by using a HPLC method.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco C Groppo, PhD, Principal Investigator — University of Campinas, Brazil; Ana PP Cione, Chem., Study Chair — BIOAGRI Laboratórios Ltda
Locations (1):
- BIOAGRI Laboratórios Ltda, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Baglie S, Rosalen PL, Franco LM, Ruenis AP, Baglie RC, Franco GC, Silva P, Groppo FC. Comparative bioavailability of 875 mg amoxicillin tablets in healthy human volunteers. Int J Clin Pharmacol Ther. 2005 Jul;43(7):350-4. doi: 10.5414/cpp43350. PMID 16035378